CLINICAL TRIAL: NCT02149511
Title: Longitudinal Morphometric Changes Following SCI
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Collaborators: Foundation Wings For Life (Other)
Responsible Party: Sponsor
Other Study IDs: KEK-ZH 2010-0271/PB_2016-00230
Record Dates: First submitted 2014-05-16; First posted 2014-05-29 (Estimated); Last update posted 2020-09-17 (Actual); Status verified 2020-08

CONDITIONS: Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- SCI subjects
- healthy control subjects

SUMMARY:
In patients with chronic spinal cord injury, imaging of the spinal cord and brain above the level of the lesion provides evidence of neural degeneration; however, the spatial and temporal patterns of progression and their relation to clinical outcomes are uncertain. New interventions targeting acute spinal cord injury have entered clinical trials but neuroimaging outcomes as responsive markers of treatment have yet to be established. We aim to use MRI to assess neuronal degeneration above and below the level of the lesion after acute spinal cord injury. In our prospective longitudinal study, we enroll patients with acute traumatic spinal cord injury and healthy controls. We assess patients clinically and by MRI at baseline, 2 months, 6 months, 12 months, and if possible 24 months and 60 months follow-up, and controls by MRI at the same timepoints. We assess cervical atrophy in white and gray matter and use cross-sectional spinal cord area measurements to assess atrophy at cervical level (C2/C3) and in the lumbar enlargement. We use myelinsensitive magnetisation transfer (MT) and longitudinal relaxation rate (R1) maps in the brain to assess microstructural changes associated with myelin. We also use diffusion tensor imaging acquired in the spinal cord at C2/C3 and in the lumbar enlargement to identify axonal loss and demyelination in the spinal white matter. Finally, we assess associations between MRI parameters and clinical improvement.

ELIGIBILITY:
Inclusion Criteria:

SCI patients:

* acute injury to the spinal cord
* no medical or mental illness
* written informed consent
* over the age of 18 years

Control subjects:

* over the age of 18 years
* written informed consent

Exclusion Criteria:

SCI patients:

* head or brain lesion associated with the trauma leading to the injury
* epileptic seizures
* MRI contraindications
* pregnant women or lactating women

Control subjects:

* pregnant women or lactating women
* MRI contraindications
* neurological or psychiatric illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Acute and chronic patients with spinal cord involvement
Sampling Method: Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2010-09; Primary Completion 2019-09 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
Cord and brain volume (mm^3) changes | Patients will be recruited within the first months of injury and scanned 6 times during the first 5 years post injury. Healthy controls will follow the same time line.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Zurich, Zurich, Switzerland